CLINICAL TRIAL: NCT05038878
Title: An Oral GnRH Antagonist to Treat Mild Autonomous Cortisol Excess (MACE) Due to Adrenal Adenomas in Postmenopausal Women
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting patients
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Alice C. Levine, Professor, Medicine - Endocrinology, Diabetes and Bone Disease, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 19-1595
Record Dates: First submitted 2021-08-17; First posted 2021-09-09 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Mild Autonomous Cortisol Excess
Keywords: mild autonomous cortisol excess (MACE); adrenal adenomas; postmenopausal women; GnRH antagonist
MeSH Terms: interventions — elagolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GnRH antagonist (Elagolix) (Experimental): Post-menopausal women with benign appearing adrenal adenomas, absence of clinical features of overt Cushing's signs or symptoms and MACE confirmed on either 24 hr urine free cortisol (UFC), late night salivary cortisol and/or abnormal dexamethasone suppression
  Interventions: Drug: Elagolix

INTERVENTIONS:
Drug: Elagolix — Patients will be given Elagolix 200 mg orally twice daily for a total of 6 months

SUMMARY:
The purpose of this research study is to determine if treatment with Elagolix will improve body weight, waist circumference, muscle strength, cortisol secretion, blood glucose, cholesterol, and bone quality as well as mood and quality of life in a female patient with mild hypercortisolism from adrenal overproduction of cortisol. Many people with adrenal nodules, or non-cancerous growths in the adrenal glands, have mildly elevated cortisol levels. Cortisol is a hormone normally made by the adrenal glands. It is increasingly being recognized that even mild elevations in cortisol levels can negatively impact blood glucose levels, serum cholesterol levels, weight and other metabolic parameters. This can lead to an increase in risk for cardiovascular disease. The study team is trying to determine if the medication Elagolix might be an effective treatment for post-menopausal females with mild hypercortisolism. Elagolix is a medication used to treat a medical condition called endometriosis by decreasing the body's production of sex hormones. Growth of adrenal adenomas is thought to be driven by such sex hormones. Therefore, by decreasing production of these hormones, the study team hopes to treat hypercortisolism caused by adrenal adenomas.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women that have incidentally found adrenal adenomas with benign appearing characteristics on imaging (<4 cm, non-contrast CT <10 HU and/or lipid rich and benign appearing on MRI)
* Absence of anti-anabolic clinical features of overt Cushing's signs (proximal muscle weakness, >three ecchymoses, hyperpigmented striae) and 2 of 3 of the following:

  * Elevated 24 hr urine free cortisol (UFC) above the upper limit of normal (>50 mcg/24 hours) in at least two complete 24-hour tests and/or
  * Late night salivary cortisol more than upper limit of normal in at least two tests and/or
  * an abnormal dexamethasone suppression defined as post 1mg dexamethasone suppression test serum cortisol concentration of >1.8 mcg/ml
* Clinic status of cessation of menses for 12 mo in a previously cycling woman and reflecting complete or nearly complete permanent cessation of ovarian function and fertility (26).
* Patients with osteoporosis that are not receiving treatment with either antiresorptive medications (bisphosphonates, denosumab) or anabolic agents (teriparitide, abaloparatide or romosozumab)

Exclusion Criteria:

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice C Levine, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Privacy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GnRH Antagonist (Elagolix)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.25 (5.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change in Cortisol Level
Description: Cortisol level after dexamethasone suppression test which measures whether adrenocorticotrophic hormone (ACTH) secretion by the pituitary can be suppressed.
  Number of participants with interval improvement and normalization of late-night salivary results after 6 months of treatment.
Time Frame: baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 4
Participants | 2

2. Primary Outcome: Change in Cortisol Level
Description: Cortisol level after dexamethasone suppression test which measures whether adrenocorticotrophic hormone (ACTH) secretion by the pituitary can be suppressed.
  Cortisol secretion as reported below by assessment of pre-treatment and post-treatment of late-night salivary cortisol levels (normal midnight values: <0.010 - 0.090)
Time Frame: baseline and 6 months
Measure: Median (Full Range); unit: ng/mL
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 4
ng/mL
  Baseline Salivary #1 | 0.252 [0.192 to 0.347]
  Baseline Salivary #2 | 0.092 [0.045 to 0.161]
  6 months Salivary #1 | 0.092 [0.053 to 0.124]
  6 months Salivary #2 | 0.4355 [0.035 to 0.78]

3. Primary Outcome: Number of Participants With Change in 24 Hour Urine Free Cortisol Level
Description: 24 hour urine free cortisol measurements. The cortisol urine test measures the level of cortisol in the urine. Cortisol is a glucocorticoid (steroid) hormone produced by the adrenal gland.
  Number of participants with improvement in 24-hour urinary free cortisol after treatment (normal 24-hr urinary cortisol is between 6 - 42 ug/24 hr).
Time Frame: Baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 4
Participants | 1

4. Primary Outcome: 24 Hour Urine Free Cortisol Level
Description: 24 hour urine free cortisol measurements. The cortisol urine test measures the level of cortisol in the urine. Cortisol is a glucocorticoid (steroid) hormone produced by the adrenal gland.
  Cortisol secretion as reported below by assessment of pre-treatment and post-treatment of 24-hour urinary cortisol levels (normal 24-hr urinary cortisol is between 6 - 42 ug/24 hr).
Time Frame: Baseline and 6 months
Measure: Median (Full Range); unit: ug/24 hour
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 4
ug/24 hour
  baseline | 14 [13 to 66]
  6 months | 23 [12 to 32]

5. Primary Outcome: Number of Participants With Change in Adenoma Size as Compared to Baseline
Description: All patients will have baseline imaging (CT or MRI) within 6 months to start of treatment and then will have repeat imaging with CT abdomen without contrast at 6 months to determine the effect of elagolix treatment on adrenal adenoma size and imaging characteristics. The images will be reviewed by a dedicated adrenal radiologist for consistency.
Time Frame: Baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 4
Participants | 0

6. Primary Outcome: Change in Adenoma Size as Compared to Baseline
Description: as for outcome 5
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 4
cm
  baseline (MRI) Right | 1.78 (0.26)
  6 months (CT) Right | 1.8 (0.22)
  baseline (MRI) Left | 2.33 (1.27)
  6 months (CT) Left | 2.13 (1.29)

7. Secondary Outcome: Change in Body Weight as Compared to Baseline
Description: Mean percent change in body weight is measured in kilograms at 6 months compared to baseline
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: percent change in body weight
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 4
percent change in body weight | 1.86 (11.4)

8. Secondary Outcome: Change in Body Weight for Those Participants Who Lost Weight
Description: Mean percent change in body weight is measured in kilograms at 6 months compared to baseline
Time Frame: baseline and 6 months
Population: Data for participants who lost weight
Measure: Mean (Standard Deviation); unit: percent change in body weight
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 3
percent change in body weight | -3.86 (0.6)

9. Secondary Outcome: Trunk Fat
Description: Trunk Fat composition assessed by DEXA scans at baseline and at 6 months.
Time Frame: baseline and 6 months
Population: Data for participants who completed dexa scan at both timepoints
Measure: Mean (Standard Deviation); unit: percent of total fat
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 2
percent of total fat
  Baseline | 44.7 (3.9)
  6 months | 42.6 (1.6)

10. Secondary Outcome: Preserved Glucose
Description: fasting blood sugar
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 4
mg/dL
  Baseline | 136.5 (51.9)
  6 months | 126.75 (41.6)

11. Secondary Outcome: Number of Participants With Vertebral Fractures
Description: Number of participants with vertebral fractures to measure rates will be assessed by lateral X-rays of thoracic and lumbar spine.
Time Frame: baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 4
Participants
  Baseline | 0
  6 months | 0

12. Secondary Outcome: The Cushing's Quality of Life Questionnaire
Description: The Cushing's Quality of Life Questionnaire is converted to a 0-100 scale in which 0 indicates the worse and 100 the best possible quality of life.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 4
score on a scale
  baseline | 70 (9.2)
  6 months | 83 (7.0)

13. Secondary Outcome: Beck's Depression Scale
Description: Beck's Depression Scale is scored on a scale of 1 to 40, where the higher score indicates severe or extreme depression.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 4
score on a scale
  baseline | 29 (10.1)
  6 months | 22 (8.3)

14. Secondary Outcome: State Trait Anxiety Inventory (STAI)
Description: The State Trait Anxiety Inventory gives a score range from 6-24 with the higher score indicating a higher level of anxiety.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GnRH Antagonist (Elagolix)
Number analyzed (Participants) | 4
score on a scale
  baseline | 17 (5.4)
  6 months | 12 (3.8)

ADVERSE EVENTS:
Time Frame: 6 months
Description: There were no adverse events.
Arm/Group | GnRH Antagonist (Elagolix)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT05038878/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT05038878/ICF_001.pdf